CLINICAL TRIAL: NCT05256212
Title: Occupational Exposure of Firefighters to Environmental Pollutants
Status: Completed | Type: Observational
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Collaborators: Ben-Gurion University of the Negev (Other)
Responsible Party: Principal Investigator, Elkana Kohn, Head of Research- Clinical Pharmacology and Toxicology, Assaf-Harofeh Medical Center
Other Study IDs: 0167-17-ASF
Record Dates: First submitted 2022-01-10; First posted 2022-02-25 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Healthy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — urine, serum, full blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- firefighters: firefighters in active service
  Interventions: Other: exposure to environmental contaminants

INTERVENTIONS:
Other: exposure to environmental contaminants — to measure levels of contaminants in different matrixes

SUMMARY:
The aim of the current trial is to assess the exposure of firefighters (FF) to environmental pollutants emitted from fires, to explore the association of exposure with their health status and to compare these data with those of non-FF participants

DETAILED DESCRIPTION:
Occupational exposure of firefighters to environmental contaminants Background Firefighters (FF) are exposed during their firefighting activities to a vast array of contaminants and toxic gases vapors that are released into the environment as results of combustion. Between those materials, there are heavy metals, brominated flame retardants (Polybrominated diphenyl ethers, PBDEs) and Volatile organic Compounds (VOC) that include between others Benzene, Toluene, Ethylbenzene and Xylene (BTEX).In the last decade a concern for negative health impact for all these contaminants appeared.

There is a vast use of these materials in the production of cars, furniture, electrical appliances, mattresses, paints, etc. These materials are released into the environment and absorbed by the human body.

There are some groups with increased exposure to these materials in comparison to the general population, as results of occupational exposure. Some of these groups include FF, workers who recycle electronic equipment and furniture manufacture workers.

Purposes:

1. to measure the levels of PBDEs, heavy metals and BTEX metabolites in the blood and urine of FF who are exposed to fires during their work
2. to evaluate the association between the levels of these materials and the health status of the participants. This will be done using a health questionnaire and the results of blood tests showing liver, renal and thyroid functions.
3. to compare their exposure levels and health status with those of general population

This is a prospective observational trial in a FF group. Exposure data from the activity log for each of the FF will also be collected.

Bromide flame retardants PBDEs

These materials are added during the manufacture process to many products such as: plastic, textile, furnitures, mattresses and electric equipment in order to reduce their flammability.

There are 5 main groups of flame retardants and more than 75 different kinds. BSEF (2006) reported the highest consumption of decaBDE at 65.7 kt in 2002, The wide manufacture and use of PBDEs increases their release and their accumulation in the environment with time.

Although PBDEs increase the safety of products in times of fire, they can release unwanted byproducts such as: dibenzene dioxinbromide and dibenzenofuran bromide.

During the last years, there is an increasing concern re. the nocive effects of these materials when they accumulate in the body.

Earlier animal studies show toxic effects of flame retardants: developmental neurotoxicity, hormonal effects and morphological renal and liver changes.

Additional studies show effects on sex hormones, ano-genital distance, puberty onset and spermatogenesis.

VOC-BTEX: these are aromatic hydrocarbon compounds, widely used in industry. They are a significant part of the air pollutants.

They have low boiling point and their main way of exposure is via the air. Humans are exposed to them from different sources: cleaning products, paints, solvents, cosmetics, car exhaust gases and cigarettes smoking.

Exposure to VOC can increase risk of congenital malformations, neuro-cognitive impairment, asthma and cancer.

During combustion, VOC are released into the environment. They may harm many systems in the body: neural, respiratory, reproductive. They also harm the liver and are mutagenic and immunotoxic.

Heavy metals (HM)

Humans are exposed to HM via the air, water or food. At high levels, all HM can harm the lungs. Some of the HM are more harmful than others:

Lead -Pb is known for neurological and cognitive harmful effects. Can also harm red blood cells, aminoacids metabolism and other metabolic systems.

Mercury -Hg can harm CNS, kidneys and embryos. Short exposure at high levels may harm: lungs, blood tension and heartbeat, digestive system, skin and eyes.

Cadmium- Cd causes abortion and preterm deliveries and can cause acidosis. Chromium-Cr: hexavalent chromium may cause skin, eyes and respiratory problems. Chronic exposure can cause cancer.

Study Plan

1. Trial population

   FF will be recruited (200). Exposure levels will be assessed for each participant by means of a detailed questionnaire. Levels of HM, PBDEs and BTEX found in blood and urine will be evaluated against health parameters such as: liver, renal and thyroid function, considering demographical , occupational and health variables (age, tenure, known diseases, eating habits, smoking and drinking.
2. Data and specimen collection

   From each FF, urine and blood (30 cc) samples will be collected and keep refrigerated till arrival into the lab. Samples will be separated and the ones for pollutants analysis will be kept in deep freezer (-80C) till analyzed.
3. Questionnaires FF will fill up specific questionnaires regarding demography, life-style, life habits during non-working hours. Basic health status, chronic diseases related to thyroid, fertility, psychological problems, both prescription and non-prescription drugs use.
4. Occupational data General data is routinely collected at the FF station such as work procedures, drills, number of calls.

   In addition, personal data will be collected for each FF: tenure, shifts/year, fire calls or other calls/year, task at the station , etc.
5. Lab tests:

Thyroid function: the following will be tested: 4-FT4; TSH; TPO-Ab Tg-Ab at Shamir MC central Lab using SOP Renal function: creatinine and GFR will be measured. Liver function: AST and ALT will be measured

PBDEs will be measured by GC-MS BTEX metabolites will be measured by LC-MS/MS Heavy Metals will be measured by ICP-MS

As a control group, samples collected in 12/12 trial (NCT03084445) that were not yet analyzed will be used. These samples were collected from men arriving to Shamir MC delivery room with their spouses.

ELIGIBILITY:
Inclusion Criteria:

* active firefighters

Exclusion Criteria:

* Women

firefighters with known liver, renal or thyroid problems

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Firefighters
Sampling Method: Non-Probability Sample
Enrollment: 108 (Actual)
Dates: Start 2017-08-15 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
PBDEs levels, measured in serum by GC-MS | Day 1- day of recruitment
  to test for PBDE levels in blood
BTEX levels, measured in urine by LC-MS/MS | Day 1- day of recruitment
  to test for BTEX levels in blood
Heavy metals (Pb, Hg, Cd) levels, measured in urine by ICP-MS | Day 1- day of recruitment
  to test for Heavy metals levels

SECONDARY OUTCOMES:
Liver enzymes levels (x2 of Upper Limit of Normal), measured in serum | Day 1- day of recruitment
  to test for liver function
renal function (eGFR<60), by creatinine level measured in serum | Day 1- day of recruitment
  to test for renal function
Thyroid function (TSH or FT4 out of lab reference values) measured in serum | Day 1- day of recruitment
  to test for thyroid function

CONTACTS AND LOCATIONS:
Overall Officials: Matityahu Berkovitch, Prof, Principal Investigator — Shamir MC
Locations (1):
- Assaf Harofeh Medical Center, Ẕerifin, Israel

IPD SHARING:
Plan to Share IPD: Yes
IPD to be shared as needed for QA purposes
Supporting Information: Study Protocol, SAP
Time Frame: from January 22 till December 2022
Access Criteria: for QA analysis of reviewers